CLINICAL TRIAL: NCT03050099
Title: Spectrometry for TIA Rapid Assessment (SpecTRA) Project: Study 1 Cohort 1A and 1B-Verification of Protein Biomarkers
Brief Title: SpecTRA; An Observational Study of the Verification of Protein Biomarkers in Transient Ischemic Attack.
Status: Completed | Type: Observational
Sponsor: Andrew Penn (Other)
Collaborators: Genome Canada (Other); Genome British Columbia (Industry); Genome Alberta (Other); Heart and Stroke Foundation of Canada (Other); Stroke Services BC (Unknown); Bruker Daltonics (Industry); LifeLabs (Unknown)
Responsible Party: Sponsor-Investigator, Andrew Penn, Principal Investigator, Vancouver Island Health Authority
Organization: Vancouver Island Health Authority (Other)
Other Study IDs: Island Health CREB 2013-023
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: TIA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human plasma collected within 24 hours of symptom onset; MRI; Holter +/- Extended Cardiac Monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild ACVS-definite: Clinical diagnosis of ACVS, and imaging positive (either DWI+ or CT/CTA+).
  Interventions: Other: Non-Interventional Study
- Mild ACVS-possible: Clinical diagnosis of ACVS, and DWI- and/or CTA-
  Interventions: Other: Non-Interventional Study
- Mimic: Clinical diagnosis of mimic and imaging negative.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — This is a non-interventional study. However, several blood samples will be taken which would not be taken as part of standard of care.

SUMMARY:
A multi-protein test using mass spectrometry (MS) for multiplexed protein quantitation is being developed. This test and the accompanying decision-aid software will provide Transient Ischemic Attack (TIA) results rapidly for a fraction of the price of neuroimaging. With guidance provided by this test, Emergency Department (ED) physicians can manage medical imaging questions such as the use of Computed Tomography Angiography (CTA) prior to ED discharge and appropriate (timely) referral to stroke clinics for consultation and follow-up care. The right patients will receive the right treatment, reduce unwarranted imaging risks and costs, and reduce the burden of stroke.

DETAILED DESCRIPTION:
This study represents an initial Verification study, in which Mass Spectrometry will be used to quantify a large number of blood proteins previously implicated in ACVS and mimic conditions in patients who are consented and enrolled in the Emergency Department within 24 hrs of symptom onset. 560 patients will be enrolled, and grouped into two cohorts (Cohort 1A: 220; and Cohort 1B: 350).

In Cohort 1A, each consented participant provides three blood samples: on arrival, 4-6 hours later, then ~24 hours after that, but no later than 32 hours from symptom onset. In cohort 1b, each patient provides only a single blood sample up to 24 hours from symptom onset.

A positive diffusion-weighted imaging (DWI) signal on Magnetic Resonance Imaging (MRI) or definite ischemia on Computed tomography (CT) or vascular occlusion on CTA will be used as proof of ischemia to classify the clinical phenotype into three groups (see below). A neurologist will adjudicate all cases according to a study defined adjudication protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 and older
2. Suspected TIA (as per <4 NIHSS; or ED physician referral to stroke clinic;
3. English speaking or translator available
4. Competent to provide consent and report symptoms
5. Provides at least one blood sample for the study within 24 hours after symptom onset

   * If three blood samples, then the patient is included in the Verification study 1 Cohort A.
   * If one blood sample, then patient is included in the Verification study 1 Cohort B.

Exclusion Criteria:

1. Stroke requiring admission to hospital based on only clinical observations (including CT scan) made before the MRI.
2. Unable to have MRI/CT
3. Subject unable to provide consent.
4. Isolated monocular blindness.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the hospital Emergency Department with symptoms suggesting mild ACVS and who are referred to the stroke service or TIA rapid access clinic by the emergency room physician.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The Development of a Protein Classifier for the Diagnosis of TIA in the Emergency Department. | 24 Hours
  141 proteins measured using multiple reaction monitoring mass spectrometry. Proteins were selected due to previous implication in stroke, TIA, migraine, other conditions that can be confused with ACVS, and other cardiovascular disturbances.

SECONDARY OUTCOMES:
The Development of a Clinical Classifier for the Diagnosis of TIA in the Emergency Department. | 24 Hours
  Clinical score calculated from standard clinical variables using our previously published formula. This score was developed to distinguish ACVS patients (who have had a recent ACVS) from Mimic (patients with symptoms that mimic those of ACVS).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Penn, M.D, Principal Investigator — Vancouver Island Health Authority; Shelagh Coutts, M.D., Principal Investigator — Alberta Health services; Christoph Borchers, P.hD, Principal Investigator — UVic- Genome BC Proteomics Centre
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver Island Health Authority, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Penn AM, Lu L, Chambers AG, Balshaw RF, Morrison JL, Votova K, Wood E, Smith DS, Lesperance M, del Zoppo GJ, Borchers CH; SpecTRA Study Group. Exploring phlebotomy technique as a pre-analytical factor in proteomic analyses by mass spectrometry. Genome. 2015 Dec;58(12):569-76. doi: 10.1139/gen-2015-0036. Epub 2015 Jul 10. PMID 26484650
- [Derived] Penn AM, Croteau NS, Votova K, Sedgwick C, Balshaw RF, Coutts SB, Penn M, Blackwood K, Bibok MB, Saly V, Hegedus J, Yu AYX, Zerna C, Klourfeld E, Lesperance ML. Systolic blood pressure as a predictor of transient ischemic attack/minor stroke in emergency department patients under age 80: a prospective cohort study. BMC Neurol. 2019 Oct 25;19(1):251. doi: 10.1186/s12883-019-1466-4. PMID 31653207